CLINICAL TRIAL: NCT04127097
Title: The Effect of Watching Cartoons During Treatment on Children's Anxiety and Fear Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Tuba Koc Ozkan, Principal Investigator, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/6-2
Record Dates: First submitted 2019-10-12; First posted 2019-10-15 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Nursing Caries; Anxiety; Fear
Keywords: anxiety; fear; nursing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cartoon group (Experimental)
  Interventions: Other: cartoon group
- control group (No Intervention)

INTERVENTIONS:
Other: cartoon group — The children in the groups were distracted by watching cartoon 2 minutes before treatment, until the process was over
  Arms: cartoon group

SUMMARY:
Objective: The study was carried out in a randomized controlled manner to determine the effect of the watching cartoons on the fear and anxiety levels of children during treatment.

Method: The population of the study consisted of children aged 5-10 years who were brought to a state hospital in a southeastern province for blood collection. A total of 92 children, 43 of whom were in the cartoon group and 49 of which were in the control group, were included in the study. Research findings; Data Form was obtained by using Child Anxiety Scale and Child Fear Scale. The children in the cartoon group were shown the cartoons they wanted during the treatment. Anxiety and fear levels before and during the blood collection were evaluated in the cartoon and control groups. The anxiety level of the children was evaluated according to their own expressions, and the level of fear was evaluated independently according to both the children's own statements and the observers' statements.

ELIGIBILITY:
Inclusion Criteria:

* being healthy
* ability to express himself/herself verbally
* having no visual or auditory problems

Exclusion Criteria:

* mental disease
* neurological disease

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Children Fear Scale | 1 minute
  The scale is used to evaluate the anxiety level of 4-10 year-old children. Five images of cartoon faces are used in the scale. Anxiety level is evaluated with numbers between "0" and "4". While "0" point refers to "no anxiety", "4" points refer to "severe anxiety"
Children Anxiety Scale | 1 minute
  it is similar to a thermometer with a bulb at the bottom and horizontal lines at upwardly spaced intervals. In the scale for children aged four to ten years, the child is asked to indicate that he / she feels "now için to measure State anxiety. Score can vary from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Batman obstetrics and pediatric hospital, Batman, Turkey (Türkiye)